CLINICAL TRIAL: NCT05819918
Title: Calcifediol in the Treatment of COVID 19. Modification of Therapeutic Response by Best Available Treatment or Other Treatment or Clinical Variables
Brief Title: Calcifediol in the Treatment of COVID 19
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: TD-CCRC-21
Record Dates: First submitted 2023-04-17; First posted 2023-04-19 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Calcifediol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calcifediol
  Interventions: Drug: Calcifediol
- Best therapy available
  Interventions: Drug: Best available therapy

INTERVENTIONS:
Drug: Calcifediol — Subjects hospitalized with COVID-19 treated with calcifediol
  Groups: Calcifediol
Drug: Best available therapy — Subjects hospitalized with COVID-19 treated with Azithromycin, hydroxychloroquine, corticoids and others authorized treatments.
  Groups: Best therapy available

SUMMARY:
Patients hospitalized with COVID-19 treated with calcifediol during the first outbreaks of the pandemic (until the first vaccinations) are compared with the aim of determining the therapeutic, clinical, functional, and biochemical variables that modify the response (admission to ICU or death) to calcifediol during hospitalization for COVID 19

DETAILED DESCRIPTION:
The ongoing pandemic of coronavirus disease-19 (COVID-19), caused by the β-coronavirus SARS-CoV-2, is the greatest challenge ever faced by modern medicine and public health systems worldwide. In early outbreaks, approximately 20% progressed to severe symptomatology, of which 5% developed acute respiratory distress syndrome (ARDS), septic shock and multi-organ failure accompanied by a high risk of death. In this scenario, the scientific community employed strong social containment measures and developed vaccines effective in preventing severe clinical forms of COVID-19. Vaccines against the causative virus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), have shown a preventive effect against the occurrence and severity of COVID-19, and social and economic activities are gradually recovering worldwide.

The rapid mutation rate of this virus family including multiple mutations in the receptor binding domain of the spike protein that have been associated with increased transmissibility and immune evasion after natural infection and vaccination, calls into question both the efficacy of vaccines and their long-term safety and the efficacy of monoclonal antibodies withdrawn for lack of effectiveness. Moreover, the cost/benefit of newly licensed oral antivirals for high-risk patients in higher-income countries remains inadequately documented.

These data update the repositioning strategy employed since the beginning of the pandemic for the use of safe drugs, approved for another indication and reproposed to improve symptoms and clinical outcomes in COVID-19 patients.

Numerous drugs have been investigated with this strategy and many studies have been published. Calcifediol (25OH vitamin D3) is one of them. Calcifediol is the prohormone of the vitamin D endocrine system (VDES). It requires hydroxylation to convert to calcitriol (1,25(OH)2 vitamin D3) , the active form that exerts its functions by activating the vitamin D receptor (VDR), which is expressed in the immune system and many other affected organs in COVID, including the lungs.

Available data strongly suggest that treatment with calcifediol can decrease the severity of COVID-19, decreasing the need for intensive care unit (ICU) admissions and decreasing the risk of mortality. It is a cost-effective treatment, without major adverse effects, and widely available, which could have positive implications for the treatment of the disease worldwide.

Another family of repositioned drugs has been the corticosteroids. Commonly used for decades for their immunosuppressive/anti-inflammatory properties by inhibiting the expression of multiple pro-inflammatory cytokines and chemokines, and the (in)activation of various immune cells. However, at the start of the pandemic in 2020, corticosteroid treatment in COVID-19 was formally contraindicated or not recommended.

Corticosteroids had been widely used during outbreaks of severe acute respiratory syndrome (SARS)-CoV and Middle East respiratory syndrome (MERS)-CoV, but review of their use in those epidemics suggested that corticosteroid use could increase mortality and secondary infection rates by delaying viral clearance. Therefore, World Health Organization (WHO) interim guidance on the clinical management of severe acute respiratory infection when SARS-CoV-2 infection was suspected (published on 28 January 2020) advised against the use of corticosteroids unless otherwise indicated.

For this reason, the three studies described that treated COVID with high-dose calcifediol and best available therapy did not use corticosteroids (except rarely and after a consensus clinical decision by the treating physicians). Thus, the results obtained did not have the confounding factor of modulation of innate and acquired immunity by corticosteroid treatment.

Following the RECOVERY trial, one of the largest randomized controlled trials for COVID-19 treatment, clinical practice guidelines were modified worldwide to authorize the standard use of dexamethasone or other corticosteroids as the best available treatment in hospitalized patients with severe COVID-19 requiring intensive oxygen therapy. However, the appropriate time interval for corticosteroid administration is a matter of debate, and the response to treatment is also likely to be related to the natural history of each patient's clinical and biological evolution. In addition, it is unclear how long treatment should last; since prolonged corticosteroid treatment may not be safe, due to interference with clotting and metabolic pathways, disease symptoms and long-term persistence of COVID-19.

Therefore, systemic glucocorticoids, included as the best available treatment, could, depending on the timing of their introduction, modify and/or confound the beneficial effect of calcifediol evidenced in the pre-corticoid stage of the pandemic. Other variables may also act as a confounding factor in the response to calcifediol treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 90 years.
* Diagnosis confirmed by positive polymerase chain reaction (PCR) for COVID-19.
* Radiological image compatible with pulmonary involvement by COVID-19.
* Admission to "Reina Sofia university Hospital (HURS)" Pneumology Department.

Exclusion Criteria:

* Patients for whom electronic medical record data cannot be collected.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients requiring hospital admission due to respiratory infection confirmed by SARS-CoV-2 (radiographic pattern of viral pneumonia and positive PCR for SARS-CoV-2) with a CURB65 severity scale (recommending hospital admission in case of a total score > 1).
  Patients meeting ALL inclusion criteria and NO exclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Need for ICU admission | from hospitalization till discharge /death
  Measure the need for ICU admission by differentiating the groups calcifediol yes/no; corticosteroids yes/no.
Mortality | from hospitalization till discharge /death
  Measure mortality by differentiating groups: calcifediol yes/no; corticosteroids yes/no.
Composite variable poor prognosis, (ICU&death) | from hospitalization till discharge /death
  Measure the composite variable poor prognosis, (ICU&death) by differentiating the groups calcifediol yes/no; corticosteroids yes/no.

SECONDARY OUTCOMES:
clinical variables that calcifediol response | from hospitalization till discharge /death
  To detect clinical variables that may modify the response to calcifediol.
drug modifying calcifediol response | from hospitalization till discharge /death
  To detect clinical variables that may modify the response to calcifediol.

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Entrenas Costa, MD, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Córdoba, Spain

REFERENCES:
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] Grana C, Ghosn L, Evrenoglou T, Jarde A, Minozzi S, Bergman H, Buckley BS, Probyn K, Villanueva G, Henschke N, Bonnet H, Assi R, Menon S, Marti M, Devane D, Mallon P, Lelievre JD, Askie LM, Kredo T, Ferrand G, Davidson M, Riveros C, Tovey D, Meerpohl JJ, Grasselli G, Rada G, Hrobjartsson A, Ravaud P, Chaimani A, Boutron I. Efficacy and safety of COVID-19 vaccines. Cochrane Database Syst Rev. 2022 Dec 7;12(12):CD015477. doi: 10.1002/14651858.CD015477. PMID 36473651
- [Background] Giliberto Capano, Michael Howlett, Darryl S L Jarvis, M Ramesh, Long-term policy impacts of the coronavirus: normalization, adaptation, and acceleration in the post-COVID state, Policy and Society, 2022; 41 (1): 1-12, doi: 10.1093/polsoc/puab018.
- [Background] Kato Y, Nishiyama K, Nishimura A, Noda T, Okabe K, Kusakabe T, Kanda Y, Nishida M. Drug repurposing for the treatment of COVID-19. J Pharmacol Sci. 2022 Jul;149(3):108-114. doi: 10.1016/j.jphs.2022.04.007. Epub 2022 Apr 25. PMID 35641023
- [Background] San Filippo S, Crovetto B, Bucek J, Nahass RG, Milano M, Brunetti L. Comparative Efficacy of Early COVID-19 Monoclonal Antibody Therapies: A Retrospective Analysis. Open Forum Infect Dis. 2022 Feb 14;9(4):ofac080. doi: 10.1093/ofid/ofac080. eCollection 2022 Apr. PMID 35299987
- [Background] Jayk Bernal A, Gomes da Silva MM, Musungaie DB, Kovalchuk E, Gonzalez A, Delos Reyes V, Martin-Quiros A, Caraco Y, Williams-Diaz A, Brown ML, Du J, Pedley A, Assaid C, Strizki J, Grobler JA, Shamsuddin HH, Tipping R, Wan H, Paschke A, Butterton JR, Johnson MG, De Anda C; MOVe-OUT Study Group. Molnupiravir for Oral Treatment of Covid-19 in Nonhospitalized Patients. N Engl J Med. 2022 Feb 10;386(6):509-520. doi: 10.1056/NEJMoa2116044. Epub 2021 Dec 16. PMID 34914868
- [Background] Reis S, Metzendorf MI, Kuehn R, Popp M, Gagyor I, Kranke P, Meybohm P, Skoetz N, Weibel S. Nirmatrelvir combined with ritonavir for preventing and treating COVID-19. Cochrane Database Syst Rev. 2022 Sep 20;9(9):CD015395. doi: 10.1002/14651858.CD015395.pub2. PMID 36126225
- [Background] Quesada-Gomez JM, Entrenas-Castillo M, Bouillon R. Vitamin D receptor stimulation to reduce acute respiratory distress syndrome (ARDS) in patients with coronavirus SARS-CoV-2 infections: Revised Ms SBMB 2020_166. J Steroid Biochem Mol Biol. 2020 Sep;202:105719. doi: 10.1016/j.jsbmb.2020.105719. Epub 2020 Jun 11. PMID 32535032
- [Background] Entrenas Castillo M, Entrenas Costa LM, Vaquero Barrios JM, Alcala Diaz JF, Lopez Miranda J, Bouillon R, Quesada Gomez JM. "Effect of calcifediol treatment and best available therapy versus best available therapy on intensive care unit admission and mortality among patients hospitalized for COVID-19: A pilot randomized clinical study". J Steroid Biochem Mol Biol. 2020 Oct;203:105751. doi: 10.1016/j.jsbmb.2020.105751. Epub 2020 Aug 29. PMID 32871238
- [Background] Nogues X, Ovejero D, Pineda-Moncusi M, Bouillon R, Arenas D, Pascual J, Ribes A, Guerri-Fernandez R, Villar-Garcia J, Rial A, Gimenez-Argente C, Cos ML, Rodriguez-Morera J, Campodarve I, Quesada-Gomez JM, Garcia-Giralt N. Calcifediol Treatment and COVID-19-Related Outcomes. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e4017-e4027. doi: 10.1210/clinem/dgab405. PMID 34097036
- [Background] Alcala-Diaz JF, Limia-Perez L, Gomez-Huelgas R, Martin-Escalante MD, Cortes-Rodriguez B, Zambrana-Garcia JL, Entrenas-Castillo M, Perez-Caballero AI, Lopez-Carmona MD, Garcia-Alegria J, Lozano Rodriguez-Mancheno A, Arenas-de Larriva MDS, Perez-Belmonte LM, Jungreis I, Bouillon R, Quesada-Gomez JM, Lopez-Miranda J. Calcifediol Treatment and Hospital Mortality Due to COVID-19: A Cohort Study. Nutrients. 2021 May 21;13(6):1760. doi: 10.3390/nu13061760. PMID 34064175
- [Background] Loucera C, Pena-Chilet M, Esteban-Medina M, Munoyerro-Muniz D, Villegas R, Lopez-Miranda J, Rodriguez-Bano J, Tunez I, Bouillon R, Dopazo J, Quesada Gomez JM. Real world evidence of calcifediol or vitamin D prescription and mortality rate of COVID-19 in a retrospective cohort of hospitalized Andalusian patients. Sci Rep. 2021 Dec 3;11(1):23380. doi: 10.1038/s41598-021-02701-5. PMID 34862422
- [Background] Shimba A, Ikuta K. Glucocorticoids Regulate Circadian Rhythm of Innate and Adaptive Immunity. Front Immunol. 2020 Sep 18;11:2143. doi: 10.3389/fimmu.2020.02143. eCollection 2020. PMID 33072078
- [Background] Dagens A, Sigfrid L, Cai E, Lipworth S, Cheng V, Harris E, Bannister P, Rigby I, Horby P. Scope, quality, and inclusivity of clinical guidelines produced early in the covid-19 pandemic: rapid review. BMJ. 2020 May 26;369:m1936. doi: 10.1136/bmj.m1936. PMID 32457027
- [Background] Stockman LJ, Bellamy R, Garner P. SARS: systematic review of treatment effects. PLoS Med. 2006 Sep;3(9):e343. doi: 10.1371/journal.pmed.0030343. PMID 16968120
- [Background] Arabi YM, Mandourah Y, Al-Hameed F, Sindi AA, Almekhlafi GA, Hussein MA, Jose J, Pinto R, Al-Omari A, Kharaba A, Almotairi A, Al Khatib K, Alraddadi B, Shalhoub S, Abdulmomen A, Qushmaq I, Mady A, Solaiman O, Al-Aithan AM, Al-Raddadi R, Ragab A, Balkhy HH, Al Harthy A, Deeb AM, Al Mutairi H, Al-Dawood A, Merson L, Hayden FG, Fowler RA; Saudi Critical Care Trial Group. Corticosteroid Therapy for Critically Ill Patients with Middle East Respiratory Syndrome. Am J Respir Crit Care Med. 2018 Mar 15;197(6):757-767. doi: 10.1164/rccm.201706-1172OC. PMID 29161116
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Sarzani R, Spannella F, Giulietti F, Di Pentima C, Giordano P, Giacometti A. Possible harm from glucocorticoid drugs misuse in the early phase of SARS-CoV-2 infection: a narrative review of the evidence. Intern Emerg Med. 2022 Mar;17(2):329-338. doi: 10.1007/s11739-021-02860-3. Epub 2021 Oct 31. PMID 34718937
- [Background] Update to living WHO guideline on drugs for covid-19. BMJ. 2021 Sep 23;374:n2219. doi: 10.1136/bmj.n2219. No abstract available. PMID 34556469
- [Derived] Blazquez-Cabrera JA, Torres-Hernandez J, Bouillon R, Casado-Diaz A, Quesada-Gomez JM, Navarro-Casado L. ALBACOVIDIOL Study: Effect of Calcifediol Treatment on Mortality in Patients Hospitalized for COVID-19: A Retrospective Analysis. Nutrients. 2025 Jun 10;17(12):1968. doi: 10.3390/nu17121968. PMID 40573079
- [Derived] Entrenas-Castillo M, Entrenas-Costa LM, Pata MP, Gamez BJ, Munoz-Corroto C, Gomez-Rebollo C, Mira-Padilla E, Bouillon R, Quesada-Gomez JM. Latent Class Analysis Reveals, in patient profiles, COVID-19-related better prognosis by calcifediol treatment than glucocorticoids. J Steroid Biochem Mol Biol. 2025 Jan;245:106609. doi: 10.1016/j.jsbmb.2024.106609. Epub 2024 Aug 31. PMID 39218235